CLINICAL TRIAL: NCT01457495
Title: Study to Assess Immunogenicity and Reactogenicity of SB Biologicals' DTPa-HBV-IPV/Hib Vaccine Given as Three-dose Primary Vaccination Course Compared to DTPa-IPV/Hib and HBV Administered Concomitantly at Separate Sites
Brief Title: Immunogenicity and Safety of DTPa-HBV-IPV/Hib Compared to DTPa-IPV/Hib and HBV Administered Concomitantly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217744/031
Record Dates: First submitted 2011-10-13; First posted 2011-10-24 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B; Diphtheria; Haemophilus Influenzae Type b (Hib); Poliomyelitis; Pertussis; Tetanus
Keywords: Infants; combined vaccine; DTPa-HBV-IPV/Hib; DTPa-IPV/Hib; safety; Immunogenicity; HBV
MeSH Terms: conditions — Hepatitis B; Diphtheria; Haemophilus Infections; Poliomyelitis; Whooping Cough; Tetanus | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (2):
- DTPa 1 Group (Experimental)
  Interventions: Biological: DTPa-HBV-IPV/Hib (Infanrix-hexa™)
- DTPa 2 Group (Active Comparator)
  Interventions: Biological: DTPa-IPV/Hib (Infanrix-IPV/Hib™); Biological: HBV (Engerix™-B)

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib (Infanrix-hexa™) — 3 doses administered intramuscularly into the right thigh at study month 0, 2 and 8
  Arms: DTPa 1 Group
Biological: DTPa-IPV/Hib (Infanrix-IPV/Hib™) — 3 doses administered intramuscularly into the right thigh at study month 0, 2 and 8
  Arms: DTPa 2 Group
Biological: HBV (Engerix™-B) — 3 doses administered intramuscularly into the left thigh at study month 0, 2 and 8
  Arms: DTPa 2 Group

SUMMARY:
This study will assess the immunogenicity of GlaxoSmithKline (GSK) Biologicals' (formerly SmithKline Beecham Biologicals') DTPa-HBV-IPV/Hib (Infanrix hexa™) vaccine compared to the separate administration of DTPa-HBV-IPV (Infanrix™ penta) and Hib (Hiberix™) vaccines administered at 3 and 5 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between 12 and 16 weeks of age at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the parents or guardians of the subject after they have been advised of the risks and benefits of the study in a language which they clearly understood, and before performance of any study procedure.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days preceding the first dose of study vaccine.
* Administration of chronic immunosuppressants or immune-modifying drugs during the study period.
* Administration of a vaccine not foreseen by the study protocol during the period starting from one month before each dose and ending one month after each dose.
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B, polio and/or Hib diseases.
* History of/or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio and/or Hib disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine, including allergic reactions to neomycin and polymyxin B.
* Major congenital defects or serious chronic illness.
* Progressive neurological disorders.
* Administration of immunoglobulins and/or any blood products since birth and during the study period.
* Acute febrile illness at the time of planned vaccination.

Ages: 12 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 312 (Actual)
Dates: Start 1998-09; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with antibody titers equal to or greater than cut-off value. | One month after the 2nd dose of the primary vaccination course (month 3)

SECONDARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines in terms of number of seropositive subjects | One month after the 2nd dose (Month 3), before and one month after the 3rd dose of the primary vaccination course (Months 8 and 9)
Immunogenicity with respect to components of the study vaccines in terms of antibody titers | One month after the 2nd dose (Month 3), before and one month after the 3rd dose of the primary vaccination course (Months 8 and 9)
Immunogenicity with respect to components of the study vaccines in terms of number of subjects with a vaccine response | One month after the 3rd dose of the primary vaccination course (Month 9)
Occurrence of solicited local symptoms | Within 4 days after each vaccination and overall
Occurrence of solicited general symptoms | Within 4 days after each vaccination and overall
Occurrence of unsolicited symptoms | Within 30 days after each vaccination, and overall
Occurrence of serious AEs | Throughout the entire study (approximately 9 months per subject) up to and including 30 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline